CLINICAL TRIAL: NCT03388242
Title: Screen and Verification of Biomarkers for Early Detection of Alzheimer's Disease
Brief Title: Protein and microRNA Markers for Early Detection of Alzheimer's Disease
Status: Withdrawn | Type: Observational
Why Stopped: The research group is too busy to do this study.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhiyi Zuo, Visiting Professor, Sun Yat-sen University
Other Study IDs: SYSEC-KY-060
Record Dates: First submitted 2017-12-19; First posted 2018-01-02 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal control people: These people are age-matched with the patients with MCI. No intervention is applied.
  Interventions: Other: No intervention
- Patients with MCI: These patients have met the criteria for diagnosing MCI. No intervention is applied.
  Interventions: Other: No intervention
- Patients with AD: These patients are diagnosed with AD. No intervention is applied.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Patients will be recruited into the study in their initial visit before patients are on any drug treatments for their AD or MCI. The study does not include use of any interventions.

SUMMARY:
Blood will be harvested from three groups of people, normal control, patients with mild cognitive impairment (MCI) and patients with Alzheimer's disease (AD), 20 people per group. The blood samples will be used to determine the difference in the expression of microRNAs and proteins. Blood samples will be harvested again at 6-month interval from patients. The combination of the microRNAs and proteins that have different expression patterns between normal control and patients with MCI will be constructed in a kit to detect the difference. This kit will be used in another set of the three groups of people to determine its sensitivity and specificity in detecting patients with MCI.

DETAILED DESCRIPTION:
As discussed above, patients' blood samples will be tested by chip to test microRNA expression and liquid chromatography-mass spectrometry to determine protein expression. The differences in microRNA and protein expression among the three groups, especially between the control and MCI, will be analyzed. This information will be used to construct a kit that can contain probes to detect a few microRNAs or proteins. This kit will be used in another set of patients to check its sensitivity and specificity. The first set of patients will also be followed up every 6 months for up to 1.5 years. Blood samples will be harvested during the follow-ups. The changes in microRNAs and proteins will be correlated with the changes of cognition. This information will be used for constructing the kit as well.

ELIGIBILITY:
Inclusion Criteria:

* Age-matched with patients with MCI group

Exclusion Criteria:

* With cognitive dysfunction
* With major cardiovascular diseases, especially stroke and brain transient ischemic attack
* On steroid treatment
* with major organ diseases

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People in general clinic or from community.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Fold changes of microRNAs in the blood of Patients with MCI over control people. | Patients with MCI and AD will be evaluated every 6 month for 1.5 years to monitor the changes in their cognition and the expression patterns of microRNAs and proteins.
  serum and plasma will be used in the screen.
Fold changes of proteins in the blood of Patients with MCI over control people. | Patients with MCI and AD will be evaluated every 6 month for 1.5 years to monitor the changes in their cognition and the expression patterns of microRNAs and proteins.
  serum and plasma will be used in the screen.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyi Zuo, MD, Ph.D., Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No
We will NOT share individual participant data with other researchers.